CLINICAL TRIAL: NCT04069182
Title: Behavioral Activation Therapy for Medical Students With Symptoms of Depression in Two Cities of Mexico
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Baja California (Other)
Collaborators: Universidad Autonoma de Ciudad Juarez (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Alejandro Dominguez Rodriguez, Full time professor of Psychology, Universidad Autonoma de Baja California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 714/2019-1
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Depression, Anxiety
Keywords: Depression; Anxiety; Medicine students
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: All the patients will be assigned to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Activation Therapy (Other): Psychological intervention
  Interventions: Behavioral: Behavioral Activation Therapy

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy — Behavioral Activation Therapy (BAT) has its origins in Cognitive Behavioral Therapy. In BAT, the patient monitors his emotions and daily activities, as a behavioral element. It seeks to increase the number of pleasant activities and increase interactions with the environment. The BAT considers positive reinforcement as the main intervention strategy. The treatment focuses on helping patients to systematically increase contact with their life's reward sources and solve their problems through procedures that focus on activation and on processes that inhibit it such as escape, avoidance behaviors and ruminant thoughts. It is a brief treatment consisting of 10 to 12 sessions spaced weekly (one hour per session), the first sessions are an explanation of the treatment and depression. Subsequent sessions are based on a collaborative work where the therapist and the patient work together to find activities that are according to the needs of the patient.

SUMMARY:
This study evaluates the effectiveness of The Behavioral Activation Protocol, a psychological treatment for the intervention of mild to moderate depression. It is compared the effectiveness of the treatment with the changes of the same participants before and after the treatment. The changes are being assessed through subjective measures such as psychometrics and objective measures such as electroencephalography.

DETAILED DESCRIPTION:
Depression is currently one of the mental health disorders that have gained relevance globally due to its constant increase in recent years. In Mexico, it is the disease that occupies the fourth position of diseases that cause disability. This disorder manifests as symptoms of physical pain when it is at high levels, resulting in a decrease in the quality of life. Other symptoms are; changes in eating, sleeping habits, and also presents comorbidity with anxiety disorders. In some cases, is presented suicidal ideation and behavior.

University students belong to the vulnerable age group, among them it has been shown that it is medical students who have symptoms of depression and are 2.45 times more likely to commit suicide compared to the general population. Medical students are a population at risk taking the characteristics of mental disorders such as depression, which can lead to abandoning studies, makes it difficult to work efficiently, and is present the deterioration of social relationships.

In the statistics on the death of doctors, between 300 and 400 doctors commit suicide each year in the United States alone (2018). In contrast, in Mexico there is no reported suicide statistics in doctors, however the data shows that the phenomenon of suicide has increased in recent years in the general population.

The patients will be treated through Behavioral Activation Therapy. Through some studies, the efficacy of the Behavioral Activation Therapy has been confirmed compared to exclusively cognitive cutting therapy. Other studies have corroborated the effectiveness of Behavioral Activation Therapy through a meta-analysis comparing this model with waiting list groups, placebo, conventional treatment and has even obtained better results with drugs treating cases of severe depression.

This study will have only one intervention group, without a control group or waiting list. The patients will be submitted to pre and post treatment. The subjective measures will be:

1. -The Center for Epidemiologic Studies - Depression (CES-D) scale.
2. - The Depression, Anxiety and Stress Scale - 21 Items (DASS-21).
3. - Pittsburgh Sleep Quality Index.
4. - The Plutchik Suicide Risk Scale

Also it is planned to measure the brain activity of the patients through an electroencephalogram, specifically the alpha and beta rhythms. To perform this measure, it will be used the EMOTIVE EPOC + of 14 channels is non-invasive, painless, low cost method Used for scientific research. The 14 channels with which the device counts. It allows to measure the cerebral areas AF3, F7, F3, FC5, T7, P7, O1, O2, P8, T8, FC6, F4, F8, AF4, based on the international system 10-20.

The intervention will be implemented in two cities in two public universities. Autonomous University of Baja California at the Faculty of Medicine and Psychology and the Autonomous University of Juarez at the Institute of Biomedical Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Currently studying medicine in one of the institutions of the 2 universities where this study will be conducted.
* Showing symptoms of depression and anxiety.

Exclusion Criteria:

* Consuming drugs
* To receive another psychological treatment in the same period of the study
* To show comorbidity with a psychiatric disorder
* Moderate to high score in the suicide scale
* Recent attempt of suicide (3 months)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in the scores of the Center for Epidemiologic Studies Depression (CES-D) scale. | 2.5 to 3 months, depending on the development of the patient and the sessions needed, ranging from 10 to 12 sessions needed, once per week.
  Center for Epidemiologic Studies Depression (CES-D) is a structured self-report scale for evaluation depression symptoms. This scale assesses the number of depression symptoms within 2 weeks. The scale consists 20 items and contains 4-point score responses (0 to 3) as the following; rarely or none of the time (less than 1 day); some of a little of the time (1-2 days); occasionally or moderate amount of time (3-4 days) and most or all of the time (5-7 days). The total possible range of scores is from 0 to 60 where ^16 is the cut-off point for this scale, and higher scores indicates more symptoms of depression. It is expected a statistical significant decrease (P < 0.05) in depression symptoms.
Change in the score of Anxiety Symptoms in the Depression Anxiety Stress Scale (DASS-21). | 2.5 to 3 months, depending on the development of the patient and the sessions needed, ranging from 10 to 12 sessions needed, once per week.
  The Depression Anxiety Stress Scale-21, is a structured self-report scale that assess the subscales of anxiety, depression and stress symptoms over the past last week. Each subscale contains seven items with responses rated on a 4-point scale (0-3) as follows; 0 Did not apply at me at all; 1 Applied to me to a considerable degree, or some of the time; 2 Applied to me to a considerable degree or a good part of time; 3 Applied to me very much or most of the time. Each subscale has a cut-off point for depression (6), anxiety (5) and stress (6). It is expected a statistical significant decrease (P < 0.05) in depression and anxiety symptoms.
Change in the score of The Pittsburgh Sleep Quality Index. | 2.5 to 3 months, depending on the development of the patient and the sessions needed, ranging from 10 to 12 sessions needed, once per week.
  This instrument assesses the quality patterns of sleep. It differentiates the "poor" and "good" sleep by measuring seven areas, where the range score of answers are from 0 to 3, the global sum of this scale can be a value between 0 to 60, and the cutoff point is "5" that indicates a "poor" sleep quality. It is expected a statistical significant increase (P < 0.05) in Sleep Quality test.
Change in the Alpha rhythm measures. | 2.5 to 3 months, depending on the development of the patient and the sessions needed, ranging from 10 to 12 sessions needed, once per week.
  Change in the alpha rhythm trough the EEG measure. The increase will be shown comparing the participants in the intervention group within their own results in the pre to post measures.

SECONDARY OUTCOMES:
Change in the Plutchik Suicide Risk Scale | 2.5 to 3 months, depending on the development of the patient and the sessions needed, ranging from 10 to 12 sessions needed, once per week.
  The Plutchik Suicide Risk Scale is a structured self-report questionnaire for evaluating suicide Risk. It consists in 15 items that assess the history of suicide attempts, ideation and suicide plans. It differentiates patients with a suicide risk from the non-suicide risk. This scale has dichotomous responses of Yes/No, and has a cut-off point of 6, where a point above the cut-off means a higher suicide risk. In this study the suicidal patients are not considering for the depression treatment although is necessary assess in depressive patients to referral to specialized treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Arenas-Landgrave, PhD, Study Chair — The National Autonomous University of Mexico; Flor Rocio Ramirez-Martinez, Phd, Study Chair — Autonomous University of Juarez; Ahmed Ali Asadi-González, PhD, Study Chair — Autonomous University of Baja California
Locations (2):
- Mexico (2):
  - Autonomous University of Juarez, Juárez, Chihuahua
  - Autonomous University of Baja California, Tijuana, Estado de Baja California

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, the informed consent is already shared in the register of clinical trials.
Supporting Information: Study Protocol, ICF
Time Frame: This data will be available approximately in june 2020 and it will be permanently available. It wil be shared in the databases of the journal where the article(s) will be published
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Ruiz Flores, L., Colín Piana, R., Corlay Noriega, I., Lara Muñoz, M., & Dueñas Tentori, H. (2007). Trastorno depresivo mayor en México: la relación entre la intensidad de la depresión, los síntomas físicos dolorosos y la calidad de vida. Salud Mental, 30 (2), 25-32.
- [Background] Tolentino JC, Schmidt SL. DSM-5 Criteria and Depression Severity: Implications for Clinical Practice. Front Psychiatry. 2018 Oct 2;9:450. doi: 10.3389/fpsyt.2018.00450. eCollection 2018. PMID 30333763
- [Background] Pacheco JP, Giacomin HT, Tam WW, Ribeiro TB, Arab C, Bezerra IM, Pinasco GC. Mental health problems among medical students in Brazil: a systematic review and meta-analysis. Braz J Psychiatry. 2017 Oct-Dec;39(4):369-378. doi: 10.1590/1516-4446-2017-2223. Epub 2017 Aug 31. PMID 28876408
- [Background] Stack S. Suicide risk among physicians: a multivariate analysis. Arch Suicide Res. 2004;8(3):287-92. doi: 10.1080/13811110490436954. PMID 16081394
- [Background] Jadoon NA, Yaqoob R, Raza A, Shehzad MA, Zeshan SC. Anxiety and depression among medical students: a cross-sectional study. J Pak Med Assoc. 2010 Aug;60(8):699-702. PMID 20726214
- [Background] Cuijpers P, van Straten A, Warmerdam L. Behavioral activation treatments of depression: a meta-analysis. Clin Psychol Rev. 2007 Apr;27(3):318-26. doi: 10.1016/j.cpr.2006.11.001. Epub 2006 Dec 19. PMID 17184887
- [Background] Barraca Mairal, J. (2010). Aplicación de la Activación Conductual en un Paciente con Sintomatología Depresiva. Clínica y Salud, 21(2), 183-197.
- [Background] Carleton RN, Thibodeau MA, Teale MJ, Welch PG, Abrams MP, Robinson T, Asmundson GJ. The center for epidemiologic studies depression scale: a review with a theoretical and empirical examination of item content and factor structure. PLoS One. 2013;8(3):e58067. doi: 10.1371/journal.pone.0058067. Epub 2013 Mar 1. PMID 23469262
- [Background] Norton PJ. Depression Anxiety and Stress Scales (DASS-21): psychometric analysis across four racial groups. Anxiety Stress Coping. 2007 Sep;20(3):253-65. doi: 10.1080/10615800701309279. PMID 17999228
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Koslowsky M, Bleich A, Greenspoon A, Wagner B, Apter A, Solomon Z. Assessing the validity of the Plutchik Suicide Risk Scale. J Psychiatr Res. 1991;25(4):155-8. doi: 10.1016/0022-3956(91)90019-7. PMID 1779413
- [Background] Goldman RI, Stern JM, Engel J Jr, Cohen MS. Simultaneous EEG and fMRI of the alpha rhythm. Neuroreport. 2002 Dec 20;13(18):2487-92. doi: 10.1097/01.wnr.0000047685.08940.d0. PMID 12499854
- See also: Mexico | Institute for Health Metrics and Evaluation — http://www.healthdata.org/mexico
- See also: Physician Suicide — https://emedicine.medscape.com/article/806779-overview
- See also: Estadística a propósito del día mundial para la prevención del suicidio (Statistics regarding the World Day for the Prevention of Suicide) — https://www.inegi.org.mx
- See also: EMOTIV EPOC — https://www.emotiv.com/epoc/

DOCUMENTS (1):
  • Informed Consent Form (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT04069182/ICF_000.pdf